CLINICAL TRIAL: NCT02398422
Title: The Listening Project at Reiss-Davis/Vista Del Mar Child and Family Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Reiss-Davis Child Study Center of Vista Del Mar (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-3268
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Auditory Perceptual Disorders; Stress Disorder
Keywords: Autonomic nervous system; Auditory processing disorder; Social behavior
MeSH Terms: conditions — Auditory Perceptual Disorders; Stress Disorders, Traumatic; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Filtered Music Intervention (Experimental): Participants will be included in all pre-intervention and post-assessment measures. Participants will receive the Listening Project Protocol intervention (filtered music). The duration of the intervention is approximately 45 minutes per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol
- Nonfiltered Music Intervention (Experimental): Participants will be included in all pre-intervention and post-assessment measures. Participants will receive the Listening Project Protocol intervention (nonfiltered music). The duration of the intervention is approximately 45 minutes per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol
- Assessment-only (No Intervention): The assessment-only group will participate in all pre- and post-intervention assessments, but will not receive the Listening Project Protocol.

INTERVENTIONS:
Behavioral: Listening Project Protocol — The filtered-music intervention will consist of listening to computer-altered acoustic stimulation, designed to modulate the frequency band of vocal music passed to the participant. The frequency characteristics of the acoustic stimulation are selected to emphasize the relative importance of specific frequencies in conveying the information embedded in human speech. Modulation of the acoustic energy within the frequencies of human voice, similar to an exaggerated vocal prosody, are hypothesized to recruit and modulate the neural regulation of the middle ear muscles and to functionally reduce sound hypersensitivities and improve auditory processing.
  The non-filtered music intervention will consist of the same music as the filtered-music intervention.
  Arms: Filtered Music Intervention; Nonfiltered Music Intervention

SUMMARY:
A research project funded by the Reiss-Davis Child Study Center of Vista Del Mar (RDCSC/VDM) will be conducted on the Vista Del Mar campus of the RDCSC/VDM to evaluate the effectiveness of the Listening Project Protocol (LPP) in children who have difficulties with autonomic and behavior regulation in the classroom. The LPP is designed as a "neural exercise" to reduce auditory hypersensitivities, to improve auditory processing of speech, and to improve behavioral state regulation. The LPP uses acoustic stimulation to exercise the neural regulation of the middle ear structures to rehabilitate and to normalize the acoustic transfer function of the middle ear structures. The current study is being conducted to evaluate efficacy and feasibility of the LPP with emotionally disturbed and learning challenged young people and will use objective measures to evaluate changes in acoustic transfer function of the middle ears structures, auditory processing skills, physiological state regulation, sensory symptoms, and academic pre and post testing.

ELIGIBILITY:
Inclusion Criteria:

* children must be between ages 6-17 years
* children must be able to read/speak in English. Parents must be able to read/speak in either English or Spanish
* children must be patients, students and/or residents at Reiss-Davis/Vista del Mar

Exclusion Criteria:

* children who wear a hearing device
* children with a history of heart disease
* children who are currently being treated for a seizure disorder
* children who are non-verbal

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in auditory hypersensitivity at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention), 2 months post-intervention
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

SECONDARY OUTCOMES:
Change from baseline in state regulation at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 2 months post-intervention
  heart rate, heart period, high-frequency heart rate variability/respiratory sinus arrhythmia
Change from baseline in auditory processing at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 2 months post-intervention
  filtered words, competing words subscales of SCAN
Change from baseline in social behavior at 1 week, and at 2 months | post-intervention (within 1 week after the intervention), 2 months post-intervention
  Listening Project Parent Questionnaire
Change from baseline in middle ear transfer function at 1 week, and at 2 months | post-intervention (within 1 week after the intervention), 2 months post-intervention
  Middle Ear Sound Absorption System (MESAS)

OTHER OUTCOMES:
Change from baseline in classroom behavior at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 2 months post-intervention
  Teacher-completed ASEBA
Change from baseline in home behavior at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 2 months post-intervention
  Caregiver-completed ASEBA

CONTACTS AND LOCATIONS:
Overall Officials: Keri J Heilman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Reiss-Davis / Vista del Mar Child and Family Services, Los Angeles, California, United States